CLINICAL TRIAL: NCT02408484
Title: Prospective, Open-label, Uncontrolled, Phase III Study to Assess the Efficacy, Safety and Pharmacokinetic of Octafibrin for On-demand Treatment of Acute Bleeding and to Prevent Bleeding During and After Surgery in Paediatric Subjects With Congenital Fibrinogen Deficiency
Brief Title: Study to Assess the Efficacy, Safety and Pharmacokinetic of Octafibrin in Paediatric Subjects With Fibrinogen Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORMA-04
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Congenital Fibrinogen Deficiency
MeSH Terms: interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octafibrin (Experimental): Plasma-derived fibrinogen concentrate
  Interventions: Biological: Octafibrin

INTERVENTIONS:
Biological: Octafibrin — Plasma-derived Fibrinogen concentrate
  Other Names: Fibrinogen concentrate

SUMMARY:
This study will assess the efficacy of Octafibrin, a fibrinogen concentrate in in the on-demand treatment of spontaneous or traumatic bleeding episodes in paediatric patients less than 12 years of age.The planned study duration is up to 5 years. The study will be considered completed when a minimum of 6 subjects (i.e., at least 3 subjects aged between 0 and <6 years and 3 subjects aged between 6 and <12 years) have at least one documented bleeding episode and when in total a minimum of 2 surgical procedures have been performed.

All patients will undergo a pharmacokinetic (PK) study after screening. This will have a duration of 14 days, after which a patient can be treated for a bleeding episode or planned surgical procedure when they occur.

ELIGIBILITY:
Inclusion Criteria:

* Aged <12 years (at the start of treatment).
* Documented diagnosis of congenital fibrinogen deficiency, expected to require on-demand treatment for bleeding or surgical prophylaxis:
* Fibrinogen deficiency manifested as afibrinogenaemia or severe hypofibrino-genaemia.
* Historical plasma fibrinogen activity of <50 mg/dL or levels below the limit of detection of the local assay method.
* Expected to have an acute bleeding episode (spontaneous or after trauma) or planning to undergo elective surgery.
* Informed consent signed by the subject's legal guardian.

Exclusion Criteria:

1. Life expectancy <6 months.
2. Bleeding disorder other than congenital fibrinogen deficiency, including dysfi-brinogenaemia.
3. Prophylactic treatment with a fibrinogen concentrate.
4. Treatment with:

   * Any fibrinogen concentrate or other fibrinogen-containing blood product within 2 weeks prior to start of treatment for the PK phase, a bleeding episode, or surgery.
   * Any coagulation-active drug (i.e., non-steroidal anti-inflammatory drugs, war-farin, coumarin derivatives, platelet aggregation inhibitors) within 1 week prior to start of the PK phase or treatment for the bleeding episode or surgery, or as a planned or expected medication during the time period from Day 1 until 24 hours (i.e., 1 day) after the last Octafibrin infusion.
5. Presence or history of:

   * Hypersensitivity to study medication.
   * Deep vein thrombosis or pulmonary embolism within 1 year prior to start of treatment for the bleeding episode or surgery.
   * Arterial thrombosis within 1 year prior to start of treatment for the bleeding episode or surgery
   * Hypersensitivity to human plasma proteins.
   * Oesophageal varicose bleeding.
   * End-stage liver disease (i.e., Child-Pugh score B or C).
6. Known positive HIV infection with a viral load >200 particles/μL or >400,000 copies/mL.
7. Polytrauma 1 year prior to start of treatment for the bleeding episode or surgery.
8. Diagnosis or suspicion of a neutralizing anti-fibrinogen inhibitor currently or any time in the past.
9. Acute or chronic medical condition which may, in the opinion of investigator, affect the conduct of the study, including subjects receiving immune-modulating drugs (other than anti-retroviral chemotherapy), such as alpha-interferon, predni-sone (equivalent to >10 mg/day), or similar drugs, at study start.
10. Treatment with IMP in another interventional clinical study currently or during the past 4 weeks.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, MD, Study Director — Octapharma
Locations (4):
- India (2):
  - St. John's Medical College Hospital, Bangalore
  - S.S Institute of Medical Science and Research Center, Davangere
- Nemazee Hospital Shiraz University of Medical Sciences, Shiraz, Iran
- Hotel De Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Octafibrin: Of the 15 patients screened,14 patients received at least one infusion of Octafibrin and were included in the study safety (SAF) and full-analysis set (FAS) populations.
  For the pharmacokinetic (PK) assessment, 13 patients received a single intravenous infusion of 70mg/kg body weight (BW) of Octafibrin. Dosage of Octafibrin when treating bleeding & surgeries was individually dosed to achieve recommended target fibrinogen plasma levels.8 patients had at least 1 bleeding episode (BE) treated with Octafibrin and constitute the first bleeding (firstBLEED) population, and 8 patients had all documented BEs treated with Octafibrin and therefore constitute the all bleeding (BLEED) population. Target fibrinogen plasma level for minor bleeding were 80-100 mg/dL; major bleeding:130-150mg/dL.
  3 patients underwent surgical interventions with at least 1 infusion of Octafibrin (SURG population). Target fibrinogen plasma level for minor surgeries: 80-100 mg/dL; major surgeries: 130-150 mg/dL.
Period: Overall Study
Arm/Group | Octafibrin
Started | 15
SAF Population (SAF = safety analysis population) | 14
FAS Population (FAS = full analysis population) | 14
PK Population (PK = pharmacokinetic population) | 13
firstBLEED Population (firstBLEED population = patients that have had at least one bleeding event treated with Octafibrin) | 8
BLEED Population (BLEED population = patients with all documented BEs treated with Octafibrin) | 8
SURG Population (SURG population = patients with surgical interventions with a least one infusion of Octafibrin) | 3
Completed | 11
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Not treated during study period | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) population defined according to the intention-to-treat principle, included the 14 patients who received at least one infusion of Octafibrin, and entered the study with a confirmed congenital fibrinogen deficiency.
Groups:
- Octafibrin: The full analysis set (FAS) population defined according to the intention-to-treat principle, included the 14 patients who received at least one infusion of Octafibrin, and entered the study with a confirmed congenital fibrinogen deficiency.
Arm/Group | Octafibrin
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 6 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4
  Race: White | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 15.7 (2.82)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 19.8 (6.93)
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 111.3 (15.37)

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Assessment of the Haemostatic Efficacy of Octafibrin in the On-demand Treatment of the First Documented Bleeding Episode of Each Patient Based on a 4-point Haemostatic Efficacy Scale
Description: The overall clinical assessment of the haemostatic efficacy of Octafibrin in treating the first documented bleeding episode (BE) of each patient. The first bleeding episode covered the time from the first Octafibrin infusion until 24 hours (i.e. 1 day) after the last infusion or the end of the treatment observation period, which ever came last.
  The investigator's overall clinical assessment of haemostatic efficacy for bleeding was based on a 4-point haemostatic efficacy scale (excellent, good, moderate or none). Excellent result was defined as immediate cessation of bleeding; 'Good' was eventual complete cessation of bleeding; 'Moderate' was incomplete cessation of bleeding and 'None' was no cessation of bleeding with alternative haemostatic intervention required.
  The IDMEAC conducted an independent adjudication of all haemostatic efficacy results and evaluated the investigator's assessments of the efficacy in the treatment of each BE.
Time Frame: First Octafibrin infusion for the treatment of a bleeding episode until 24 hours (i.e., 1 day) after the last infusion or the end of the treatment observation period, whichever comes last
Population: The analysis was performed in the firstBLEED population which included patients in the full-analysis (FAS) population who had at least one bleeding episode treated with Octafibrin (n=8).
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Assessment: Efficacy rating on a 4-point efficacy scale as assessed by the Investigator
- IDMEAC Assessment: Efficacy rating on a 4-point efficacy scale as assessed by the IDMEAC
Arm/Group | Investigator Assessment | IDMEAC Assessment
Number analyzed (Participants) | 8 | 8
Participants
  Excellent | 5 | 6
  Good | 1 | 2
  Moderate | 1 | 0
  None | 1 | 0

2. Primary Outcome: Overall Clinical Assessment of the Haemostatic Efficacy of Octafibrin in the On-demand Treatment of the First Documented Bleeding Episode of Each Patient Based on a 2-point Haemostatic Efficacy Scale
Description: The overall clinical assessment of the haemostatic efficacy of Octafibrin in treating the first documented bleeding episode (BE) of each patient. The first bleeding episode covered the time from the first Octafibrin infusion until 24 hours (i.e. 1 day) after the last infusion or the end of the treatment observation period, which ever came last.
  The investigator's overall clinical assessment of haemostatic efficacy for bleeding was based on a 2-point haemostatic efficacy scale (success and failure). Efficacy rating of excellent or good on the four-point scale (above) indicated success and efficacy rating of moderate or none indicated failure.
  The IDMEAC conducted an independent adjudication of all haemostatic efficacy results and evaluated the investigator's assessments of the efficacy in the treatment of each BE.
Time Frame: From the first Octafibrin infusion until 24 hours (i.e. 1 day) after the last infusion or the end of the treatment observation period, which ever came last.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Assessment: Efficacy rating on a 2-point efficacy scale as assessed by the Investigator
- IDMEAC Assessment: Efficacy rating on a 2-point efficacy scale as assessed by the IDMEAC
Arm/Group | Investigator Assessment | IDMEAC Assessment
Number analyzed (Participants) | 8 | 8
Participants
  Success | 6 | 8
  Failure | 2 | 0

3. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Area Under the Concentration-time Curve Normalised (AUCnorm)
Description: AUCnorm (Area under the concentration-time curve normalized to the dose administered) was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: The analysis was performed in the pharmacokinetic (PK) population which included all patients in the full-analysis (FAS) population who underwent PK assessment and had at least one valid post-baseline fibrinogen activity level (n=13).
Measure: Mean (Standard Deviation); unit: h*kg*g/L/mg
Groups:
- Octafibrin: PK population
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
h*kg*g/L/mg | 1.419 (0.4385)

4. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Response - Incremental in Vivo Recovery (IVR)
Description: IVR was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Between the pre-infusion and the 3-hour post-infusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL/(mg/kg)
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
mg/dL/(mg/kg) | 1.592 (0.3224)

5. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Terminal Elimination Half-life (t1/2)
Description: t1/2 was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: The analysis was performed in the pharmacokinetic (PK) population, which included all patients in the full-analysis (FAS) population who underwent PK assessment and had at least one valid post-baseline fibrinogen activity level (n=13).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
hours | 84.356 (34.2658)

6. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Maximum Plasma Concentration (Cmax)
Description: Cmax was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: The analysis was performed in the pharmacokinetic (PK) population, which included all patients in the full-analysis (FAS) population who underwent PK assessment and had at least one valid post-baseline fibrinogen activity level.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
g/L | 1.559 (0.3183)

7. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
hours | 1.154 (0.5547)

8. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Mean Residence Time (MRT)
Description: MRT was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
hours | 114.332 (37.9732)

9. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Volume of Distribution (Vss)
Description: Vss was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
mL/kg | 81.651 (15.2735)

10. Secondary Outcome: Single-dose Pharmacokinetics of Octafibrin: Clearance (Cl)
Description: Cl was assessed after a single intravenous infusion of 70 mg/kg body weight of Octafibrin.
Time Frame: Before first infusion, 1 hour, 3 hours, 1 day, 2 days, 4 days, 7 days, 10 days and 14 days post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Octafibrin
Number analyzed (Participants) | 13
mL/h/kg | 0.756 (0.1872)

11. Secondary Outcome: Change in Maximum Clot Firmness (MCF) for the First Bleeding Episode for Each Patients and for All Bleeding Episodes
Description: MCF was measured using thromboelastometry (ROTEM). ROTEM is a method for the continuous measurement of clot formation and clot firmness. It utilises a mechanical detection system which is based on the ability of the blood or plasma clot to form a mechanical coupling over a distance of 1 mm.
  ROTEM was used to measure MCF as a surrogate efficacy marker for haemostatic efficacy before and after the first infusion of Octafibrin for treatment of the first bleeding episode and all bleeding episodes. The change in MCF was measured from baseline to 1 hour post-infusion of Octafibrin administration.
Time Frame: Before first infusion and 1 hour post-infusion of Octafibrin
Population: The analysis was performed in patients in the full-analysis set population that had at least one bleeding episode (BE) treated with Octafibrin (firstBLEED population: n=8), and all patients that had all documented BEs treated with Octafibrin (BLEED population: n=8)
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Units Other Than Participants: Number of bleeding episodes
Groups:
- Change in MCF for the firstBLEED Population: Change in MCF specifically for the first infusions of Octafibrin administered for the treatment of the first bleeding episode of the patients in the firstBLEED population.
- Change in MCF for the BLEED Population: Change in MCF for the first infusions of Octafibrin administered for the treatment of all bleeding episodes of patients in the BLEED population.
Arm/Group | Change in MCF for the firstBLEED Population | Change in MCF for the BLEED Population
Number analyzed (Participants) | 8 | 8
Number analyzed (Number of bleeding episodes) | 8 | 10
millimeter (mm) | 3.1 (1.96) | 3.3 (1.77)
Statistical Analysis 1: Comparison: Change in MCF for the firstBLEED Population; Test type: Other; p = 0.0028, ANOVA — p-value for the change in MCF from baseline to 1 hour post infusion for the firstBLEED population
Statistical Analysis 2: Comparison: Change in MCF for the BLEED Population; Test type: Other; p = 0.0002, ANOVA — p-value for the change in MCF from baseline to 1 hour post infusion for the BLEED population

12. Secondary Outcome: Change in the Fibrinogen Level for All Bleeding Episodes up to 1 Hour-post Infusion for the First Bleeding Episode and All Bleeding Episodes
Description: Change in fibrinogen level was assessed using the Clauss fibrinogen assay for the first bleeding episode and all bleeding episodes. The change in fibrinogen level was assessed from Day 1 pre-infusion to 1 hour post-infusion of Octafibrin.
Time Frame: Pre-infusion and 1 hour post-infusion of Octafibrin
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: fibrinogen level (mg/dL)
Groups:
- Change in Fibrinogen Level for the firstBLEED Population: Change in fibrinogen level specifically for the first infusions of Octafibrin administered for the treatment of the first bleeding episode of the patients in the firstBLEED population.
- Change in Fibrinogen Level for the BLEED Population: Change in fibrinogen level for the first infusions of Octafibrin administered for the treatment of all bleeding episodes of patients in the BLEED population.
Arm/Group | Change in Fibrinogen Level for the firstBLEED Population | Change in Fibrinogen Level for the BLEED Population
Number analyzed (Participants) | 8 | 8
fibrinogen level (mg/dL) | 98.9 (13.56) | 98.1 (13.33)

13. Secondary Outcome: Incremental in Vivo Recovery Following the First Infusion of Octafibrin Administration for the Treatment of the First Bleeding Episode and of All Bleeding Episodes
Description: Incremental IVR calculated as the maximum increase in plasma fibrinogen (i.e. Clauss data) between the pre-infusion and the 3-hour post-infusion measurement, (expressed as absolute concentration in plasma [mg/dL]), divided by the exact dose of Octafibrin per body weight (expressed as mg/kg dosed).
  Incremental (response) IVR data for the firstBLEED and BLEED populations were calculated.
Time Frame: Pre-infusion and 3 hours post-infusion
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: (mg/dL)/(mg/kg)
Groups:
- Incremental IVR Response for the firstBLEED Population: Incremental IVR response for the first infusions of Octafibrin administered for the treatment of the first bleeding episode of the patients in the firstBLEED population.
- Incremental IVR Response for the BLEED Population: Incremental IVR response for the first infusions of Octafibrin administered for the treatment of all bleeding episodes of patients in the BLEED population.
Arm/Group | Incremental IVR Response for the firstBLEED Population | Incremental IVR Response for the BLEED Population
Number analyzed (Participants) | 8 | 8
(mg/dL)/(mg/kg) | 1.5 (0.29) | 1.5 (0.34)

14. Secondary Outcome: Efficacy of Octafibrin in All Bleeding Episodes Based on a Four-point Haemostatic Efficacy Scale
Description: The haemostatic efficacy of Octafibrin in the on-demand treatment of all bleeding episodes was based on a 4-point haemostatic efficacy scale ranging from excellent, good moderate and none. The efficacy assessment of each patients was assessed by the Investigator and the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC).
  .
Time Frame: as for outcome 1
Population: The analysis was performed in patients in the full-analysis set population that had all documented bleeding episodes treated with Octafibrin (BLEED population: n=8)
Measure: Count of Units; unit: Number of bleeding episodes
Units Other Than Participants: Number of bleeding episodes
Groups:
- Investigator: Efficacy assessment for the treatment of all bleeding episodes according to the Investigator
- IDMEAC: Efficacy assessment for the treatment of all bleeding episode according to the IDMEAC
Arm/Group | Investigator | IDMEAC
Number analyzed (Participants) | 8 | 8
Number analyzed (Number of bleeding episodes) | 10 | 10
Number of bleeding episodes
  Excellent | 7 | 8
  Good | 1 | 2
  Moderate | 1 | 0
  None | 1 | 0

15. Secondary Outcome: Efficacy of Octafibrin in All Bleeding Episodes Based on a Two-point Haemostatic Efficacy Scale
Description: The haemostatic efficacy of Octafibrin in the on-demand treatment of all bleeding episodes was based on a 2-point haemostatic efficacy scale ranging from success to failure. The efficacy assessment of each patients was assessed by the Investigator and the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC).
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Count of Units; unit: Number of bleeding episodes
Units Other Than Participants: Number of bleeding episodes
Arm/Group | Investigator | IDMEAC
Number analyzed (Participants) | 8 | 8
Number analyzed (Number of bleeding episodes) | 10 | 10
Number of bleeding episodes
  Success | 8 | 10
  Failure | 2 | 0

16. Secondary Outcome: Efficacy of Octafibrin in Surgical Prophylaxis Based on a Four-point Haemostatic Efficacy Scale
Description: The haemostatic efficacy of Octafibrin was assessed during surgery prophylaxis by the surgeon and the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC), on a 4-point scale ranging from excellent, good, moderate and none. Intra-operative blood loss lower or equal to the average expected blood loss was rates as 'Excellent'; intra-operative blood loss higher than average expected blood loss but lower or equal to maximal expected blood loss was rated as 'Good'; intra-operative blood loss was higher than expected blood loss was rated as 'Moderate' and haemostasis that was uncontrolled and necessitated a change in clotting factor replacement regimen was rated as 'None'.
  The surgical observation period started lasted from the first dose of Octafibrin to at least 3 post-operative days for minor and 7 post-operative days for major surgeries or until the day of the last post-operative infusion, whichever comes last.
Time Frame: First dose of Octafibrin prior to surgery until last day of post-operative infusion
Population: The analysis was performed in patients in the full-analysis set population with documented surgical interventions treated with at least one infusion of Octafibrin (n=3).
Measure: Count of Units; unit: Number of surgeries
Units Other Than Participants: Number of surgeries
Groups:
- Surgeon: Intra-operative assessment of Octafibrin efficacy in surgical prophylaxis as assessed by the Surgeon.
- IDMEAC: Intra-operative assessment of Octafibrin efficacy in surgical prophylaxis as assessed by the IDMEAC.
Arm/Group | Surgeon | IDMEAC
Number analyzed (Participants) | 3 | 3
Number analyzed (Number of surgeries) | 3 | 3
Number of surgeries
  Excellent | 3 | 3
  Good | 0 | 0
  Moderate | 0 | 0
  None | 0 | 0

17. Secondary Outcome: Efficacy of Octafibrin in Surgical Prophylaxis Based on a Two-point Haemostatic Efficacy Scale
Description: The haemostatic efficacy of Octafibrin was assessed during surgery prophylaxis by the surgeon and the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC), on a 2-point scale ranging from success to failure.
  Efficacy rating of excellent or good from the 2-point efficacy scale indicated 'Success', and efficacy rating of moderate or none indicated 'Failure'.
  The surgical observation period started lasted from the first dose of Octafibrin to at least 3 post-operative days for minor and 7 post-operative days for major surgeries or until the day of the last post-operative infusion, whichever comes last.
Time Frame: First dose of Octafibrin prior to surgery until last day of post-operative infusion
Population: as for outcome 16
Measure: Count of Units; unit: Number of surgeries
Units Other Than Participants: Number of surgeries
Arm/Group | Surgeon | IDMEAC
Number analyzed (Participants) | 3 | 3
Number analyzed (Number of surgeries) | 3 | 3
Number of surgeries
  Success | 3 | 3
  Failure | 0 | 0

18. Secondary Outcome: Patients With Elevated Values of Prothrombin Fragments 1+2
Description: Thrombogenicity was assessed by measuring the plasma levels of prothrombin fragment 1 (F1) and prothrombin fragment 2 (F2), before and after each Octafibrin infusion for the treatment of bleeding episodes during the study. This outcome measure examined the number of patients with elevated values of prothrombin fragments F1 + F2 that were outside of the reference range of 69 to 229 pmol/L, three hours post-infusion with Octafibrin.
Time Frame: 3 hours post-infusion of Octafibrin
Population: The analysis was performed in all patients in the safety population that met the study inclusion criteria and received at least one infusion of Octafibrin (n=14).
Measure: Count of Participants; unit: Participants
Groups:
- Prothrombin Fragments (1+2): Patients with elevated values of prothrombin Fragments 1+2 (outside of the reference range of 69 to 229 pmol/L) 3 hours post-infusion
Arm/Group | Prothrombin Fragments (1+2)
Number analyzed (Participants) | 14
Participants | 3

19. Secondary Outcome: Safety Assessment: Immunogenicity Testing for Anti-fibrinogen Antibodies
Description: The number of patients developing anti-fibrinogen antibodies were observed during the observation period using an experimental non-standard ELISA quantitative laboratory test.
  Immunogenicity testing for the presence of anti-fibrinogen antibodies before the first infusion of Octafibrin and on Day 30 after the treatment of each bleeding episode.
Time Frame: Start of the first Octafibrin infusion to the end of each 30-day observation and follow-up period for on-demand treatment
Population: The analysis was performed in all patients in the safety population that met the inclusion criteria and received at least one infusion of Octafibrin during the study (n=14)
Measure: Count of Participants; unit: Participants
Groups:
- Octafibrin: The safety population consists of all patients that met the inclusion criteria and received at least one infusion of Octafibrin (n=14)
Arm/Group | Octafibrin
Number analyzed (Participants) | 14
Participants | 2

20. Secondary Outcome: Safety Assessment: Adverse Events
Description: Adverse events, including thromboembolic complications and early signs of allergic or hypersensitivity reactions.
Time Frame: Start of the first Octafibrin infusion to the end of PK, end of 30-day observation and follow-up period for on-demand treatment, or the end of the surgical observation period
Population: as for outcome 19
Measure: Number; unit: Number of adverse events
Arm/Group | Octafibrin
Number analyzed (Participants) | 14
Number of adverse events | 10

ADVERSE EVENTS:
Time Frame: Between the start of the first Octafibrin infusion and the end of each 30-day observation and follow-up period or during the surgical observation period, and were absent prior to treatment or worsened relative to the pre-treatment state.
Arm/Group | Octafibrin
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octafibrin (N=14)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octafibrin (N=14)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (3)
Influenza-like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT02408484/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02408484/SAP_003.pdf